CLINICAL TRIAL: NCT01557127
Title: Nexavar Dose Evaluation Study in Patients With Advanced Renal Cell Carcinoma
Brief Title: Nexavar Dosing in Renal Cancer Patients in "Real-life" Setting
Acronym: NEXST
Status: Completed | Type: Observational
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Other Study IDs: 16268
Record Dates: First submitted 2012-03-16; First posted 2012-03-19 (Estimated); Last update posted 2017-03-28 (Actual); Status verified 2017-03

CONDITIONS: Carcinoma, Renal Cell
Keywords: Renal cell carcinoma,; Sorafenib; Dosing
MeSH Terms: conditions — Carcinoma, Renal Cell | interventions — Sorafenib

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Group 1
  Interventions: Drug: Sorafenib (Nexavar, BAY43-9006)

INTERVENTIONS:
Drug: Sorafenib (Nexavar, BAY43-9006) — Patients scheduled for treatment with sorafenib given in regular daily dose i.e. 800mg (400mg bid)

SUMMARY:
This study is a registry of renal cancer patients treated with Nexavar. It aims to evaluate the actual dosing of Nexavar in "real-life" setting vs. the prescribed dose.

ELIGIBILITY:
Inclusion Criteria:

* Age >/= 18 years
* Diagnosis of renal cell carcinoma
* Failure of prior therapy with interferon-alfa (IFN) or interleukine-2 (IL-2) or disqualified from therapy with IFN/IL-2
* Patients in whom the oncologist has decide to start therapy with sorafenib.

Exclusion Criteria:

* Synonymous with contraindications to Nexavar.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with renal cell carcinoma scheduled to treatment with sorafenib, following therapy failure with IFN/IL-2
Sampling Method: Probability Sample
Enrollment: 205 (Actual)
Dates: Start 2011-11-01 (Actual); Primary Completion 2014-05-16 (Actual); Study Completion 2016-03-31 (Actual)

PRIMARY OUTCOMES:
Percentage of patients in whom the actual dose of sorafenib equaled the planned dose | 12 months

SECONDARY OUTCOMES:
Overall tolerability of treatment as measured by rate of adverse events | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- Many Locations, Poland

IPD SHARING:
Plan to Share IPD: No